CLINICAL TRIAL: NCT04600908
Title: Incidence of Commuting Accidents Among Non-physician Staff of a Large University Hospital Center From 2012 to 2016
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 07-3
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Accident, Traffic
Keywords: Commuting accident; Traffic accident; Hospital; Descriptive study; Incidence; Health care worker

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-physician staff: All non-physician staff who have had commuting accidents
  Interventions: Other: Characteristics of accidents

INTERVENTIONS:
Other: Characteristics of accidents — informations about commuting accidents were recorded either during an occupational medicine consultation or by the medical service after reception of the medical certificate and the administrative declaration

SUMMARY:
Over the past thirty years, risk of road traffic accidents has decreased but remains high and accounts for 44% of fatal work-related accidents for commuting and mission-related accidents. The aims of this study were to estimate the overall incidence of commuting accidents for non-physician professionals in a major university hospital and by gender and different professional categories, and to assess its evolution over a 5-year period. A descriptive analysis was performed on 390 commuting accidents from 2012 to 2016 extracted from the university hospital's occupational health service.

ELIGIBILITY:
Inclusion Criteria:

* non-physician staff
* commuting accidents

Exclusion Criteria:

* work accidents
* on-duty road accidents
* physician staff

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: non-physician staff working at the Hospices Civils de Lyon and having had commuting accidents between 2012 and 2016
Sampling Method: Non-Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Incidence of commuting accidents | at the enrollment
  Incidence of commuting accidents according to sex, occupational categories and year of accident.
  The evolution of the number of accidents over the years was assessed by the Cochran-Armitage Chi² trend test. Crude Relative risk (RR) and 95% confidence intervals for the association of commuting accident with respectively sex, occupational categories and years were estimated on log-binomial regression using the using the GENMOD procedure in the SAS statistical package (version 9.4) with the DIST=BINOMIAL and LINK=LOG options.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Bron, France